CLINICAL TRIAL: NCT05727462
Title: Effects of a Protocol of Soft Tissue Mobilization Techniques With or Without TECAR Treatment on Pain, Local Sensitivity, Neck Range of Motion, and Functional Ability in Woman With Chronic Neck Pain: A Randomized Clinical Trial
Brief Title: Effects of Manual Therapy With TECAR in Woman With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras PT, PhD, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-03/2023
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Neck Pain
Keywords: Neck Pain; Myofascial trigger points; Manual Therapy; TECAR; Physiotherapy
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: An assessor-blind randomized controlled trial lasting five weeks, with a six-month follow-up, will be conducted on 80 adult women with chronic neck pain and at least one trigger point in the upper trapezius muscle. Participants will be randomly allocated into two groups of 40 each (intervention and control). The intervention group will receive a combined treatment of manual techniques with two TECAR anti-static electrode bracelets, while the control group will follow the same protocol without the electrode bracelets. All participants will undergo a total of 15 treatments over the five-week period.
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy with TECAR (Experimental): Participants allocated to this group received 15 sessions of a manual therapy protocol applied by two resistive TECAR bracelet electrodes (one in each hand).
  Interventions: Other: Manual Therapy with TECAR
- Manual Therapy without TECAR bracelet electrodes (Active Comparator): Participants allocated to this group received the same Manual Therapy protocol without the resistive TECAR bracelet electrodes
  Interventions: Other: Manual Therapy without TECAR

INTERVENTIONS:
Other: Manual Therapy with TECAR — The following myofascial release techniques will be applied:
  Myofascial release of the upper trapezius Gross stretch, vertical gross stretch, and focused stretch of the upper trapezius Myofascial release at the cranial base Gross release of the sternocleidomastoid muscle
  Additionally, the following ischemic compression technique will be applied:
  Ischemic compression on the upper trapezius muscle Manual therapy manipulations will be administered in combination with a capacitive conventional electrode and two special electrode bracelets that turn the therapist's hands into anti-static electrodes. High-frequency currents will be applied at frequencies of 300 kHz, 500 kHz, and 1 MHz, with a flexible self-adhesive grounding electrode placed on the thoracic spine for reference.
  Arms: Manual Therapy with TECAR
Other: Manual Therapy without TECAR — Participants in this group will follow the same manual protocol as the first group, without the application of high-frequency current. Each manual therapy session will begin with a ten-minute preparation involving light massage and stretching. The massage will include the effleurage technique, followed by petrissage and kneading, focusing on the cervical and thoracic areas, particularly the upper trapezius, suboccipital region, and cervical paraspinal muscles. Stretching will be applied to the upper trapezius, levator scapulae, and sternocleidomastoid muscles.
  Arms: Manual Therapy without TECAR bracelet electrodes

SUMMARY:
The aim of our clinical study is to investigate the efficacy of combining a program of manual techniques for treating chronic neck pain with the simultaneous application of TECAR therapy, utilizing two specialized anti-static electrode bracelets. A total of 80 women with upper trapezius trigger points and neck pain persisting for more than 12 weeks will be randomly assigned to two groups. In the first group, combined treatment involving manual techniques and two TECAR anti-static electrode bracelets will be administered, while in the second group, the same protocol will be followed without the electrode bracelets. All participants will receive a total of 15 treatments over five weeks, with a follow-up assessment six months post-treatment. Pain will be measured using the Numerical Pain Rating Scale (NPRS), and pain thresholds at the upper trapezius muscle and suboccipital area will be evaluated with a digital algometer. Additionally, neck range of motion will be assessed with a goniometer, and functional ability will be evaluated using the "Neck Disability Index" questionnaire. Assessments will be conducted before and after the treatment period, with a follow-up assessment six months later. For statistical analysis, a multivariate analysis of variance (MANOVA) with repeated measures will be applied, with the significance level set at p < .05.

DETAILED DESCRIPTION:
Background: Chronic neck pain is defined as neck pain lasting more than 12 weeks and is often accompanied by painful trigger points in the neck muscles. The use of manual techniques, such as myofascial release and ischemic compression on painful points in the neck muscles, has been shown to reduce pain and improve functional ability and neck range of motion in individuals with chronic neck pain.

Aim: The aim of our clinical study is to investigate the efficacy of combining a program of manual techniques for treating chronic neck pain with the simultaneous application of TECAR therapy using two specialized anti-static electrode bracelets.

Method: Eighty women with upper trapezius trigger points and neck pain symptoms persisting for more than 12 weeks will be randomly assigned to two groups. The first group will receive a combined treatment of manual techniques with two TECAR anti-static electrode bracelets, while the second group will follow the same protocol without the electrode bracelets. All participants will undergo a total of 15 treatments over five weeks, with a follow-up assessment after six months. Pain will be measured using the Numerical Pain Rating Scale (NPRS), pressure pain threshold (PPT) of the upper trapezius muscle and suboccipital area will be evaluated with a digital algometer, neck range of motion (ROM) will be assessed using a goniometer, and functional ability will be measured with the "Neck Disability Index" questionnaire. Assessments will be conducted before and after the treatment period, with a follow-up assessment six months later. For statistical analysis, a multivariate analysis of variance (MANOVA) with repeated measures will be applied, with the significance level set at p < .05.

Expected Results: Modern TECAR devices, through special resistive bracelet electrodes, allow the therapist's hand to function as a mobile electrode. This enables the simultaneous effect of both therapeutic modalities-manual techniques and high-frequency current. Therefore, we expect the combination to be more effective than manual techniques alone in improving the clinical profile of adult women with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

Women with chronic neck pain lasting at least three months Presence of at least one active or latent trigger point in the upper trapezius muscle Numerical Rating Pain Scale score greater than 3 Written consent to participate in the study

Exclusion Criteria:

Participation in any form of treatment in the past three months (e.g., physiotherapy, massage, local anesthetic injections) History of neck trauma and/or surgery in the neck region Paresthesia in the neck area Implanted pacemaker Cancer Pregnancy Systemic musculoskeletal diseases, diagnosed neurodegenerative diseases (e.g., Parkinson's disease), epilepsy, or history of psychiatric disorders

Ages: 22 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity with Numeric Pain Rating Scale (NPRS) | pre-treatment, week 5, 6-month follow-up
  This tool is an eleven-point pain scale numbered from zero to 10. The left end of the scale corresponds to zero and is marked as "No pain", whereas the right end corresponds to 10 and is marked as "Maximum pain". Consequently, a higher value indicates more intense pain (Childs et al, 2005). The examinee is asked to choose an integer that best reflects the intensity of their pain. The NPRS is widely used to measure pain in both clinical practice and research, showing high test-retest reliability and high conceptual construct validity
Changes in Pressure Pain Threshold (PPT) with pressure algometry | pre-treatment, week 5, 6-month follow-up
  Pressure pain threshold (PPT) is defined as the minimum amount of pressure that induces pain. PPT was assessed using a digital algometer. Measurements were taken over the upper border of the trapezius muscle, midway between the midline and the lateral border of the acromion, as well as in the suboccipital area, 2 cm lateral to the spinous process of the axis. The metal rod of the algometer was positioned vertically on each site, and the examiner applied gradually increasing pressure at a rate of 1 kg/s. PPT was recorded in kg/cm².
Changes in functional capacity with the Greek Version of Neck disability index questionnaire | pre-treatment, week 5, 6-month follow-up
  It is a self-reported, ten-item scale, with each item assessing different aspects of neck pain complaints. Most items relate to restrictions in activities of daily living, and each item is rated on a scale of 0 to 5, where 0 indicates no disability and 5 indicates maximum disability. The total score ranges from 0 to 50. The Neck Disability Index (NDI) is well-supported in the literature and is the most commonly used tool for reporting neck pain.
Changes in Cervical Range of Motion through goniometry | pre-treatment, week 5, 6-month follow-up
  Active cervical range of motion was measured using two types of goniometers: two bubble inclinometers and a large-scale universal goniometer. Measurements included active cervical flexion, extension, rotation, and side bending, with participants seated in an upright position. Range of motion was recorded in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Paris Iakovidis, Ph.D, Study Chair — Department of Physiotherapy, International Hellenic University
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic University, Thessaloniki, Sindos Thessaloníki, Greece